CLINICAL TRIAL: NCT03323619
Title: Impact of Anesthesia Technique on Post-operative Delirium After Transcatheter Aortic Valve Implantation
Acronym: DELIRIUMTAVI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: PSS2017/DELIRIUMTAVI-MATTEI/YB
Record Dates: First submitted 2017-10-24; First posted 2017-10-27 (Actual); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Delirium; Post-Op Complication; Anesthesia; Aortic Valve Disease
Keywords: Transcatheter aortic valve replacement; Anesthesia technique; Delirium
MeSH Terms: conditions — Delirium; Postoperative Complications; Aortic Valve Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- GA: No intervention. General anesthesia is decided by the physicien according to his usual practice
  Interventions: Procedure: anesthesia type
- LASed: No intervention. Local anesthesia with sedation is decided by the physicien according to his usual practice
  Interventions: Procedure: anesthesia type

INTERVENTIONS:
Procedure: anesthesia type — No intervention. General anesthesia or local anesthesia with sedation are decided by the physicien according to his usual practice

SUMMARY:
Aortic stenosis is a frequent valvulopathy in Europe and North America. It occurs mainly over 65 years (2-7% of the population over 65 years). Treatment of symptomatic stenosis is an indication of aortic valve replacement. For patients with high surgical risk (EuroSCORE II> 6), TAVI (Transcatheter Aortic Valve Implantation) is recommended. This type of procedure concerns elderly patients (75-80 years on average in the literature) therefore the anesthesia technique must be optimal. The postoperative complications are, on the one hand, well-described surgical complications (Cardiogenic shock, bleeding, rhythm disorders, renal insufficiency) and, on the other hand, those related to anesthesia which are less well characterized. There is no consensus on best anesthesia technique for TAVI procedure managment. Between teams practices are different. It may consist of general anesthesia (GA) or local anesthesia with sedation (LASed). Elderly anesthesia has specific complications, including acute cerebral disturbances (delirium) usually occurring within 24 to 48 hours postoperatively and up to 7 days. It is recommended to screen delirium for patients admitted in intensive care using the CAM-ICU scale. The aim of the study is to observe the impact of the anesthesia technique (GA versus LASed) on delirium in post-operative aortic valve replacement with TAVI procedure

ELIGIBILITY:
Inclusion Criteria:

* Hospital admission for TAVI femoral way
* Age > 18 years
* Psychiatric disease

Exclusion Criteria:

* Opposition of the operator (Interventional Cardiologist or Surgeon) to one of the two anesthesia technique
* Contraindication to local anesthesia with sedation: agitation, delirium, allergy to local anesthetics, risk of inhalation
* Opposition of the patient to use his data for research

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patient admitted for TAVI intervention
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-11-02 (Actual); Primary Completion 2020-08-02 (Estimated); Study Completion 2020-11-02 (Estimated)

PRIMARY OUTCOMES:
Delirium | 7 days
  post-operative delirium after TAVI

SECONDARY OUTCOMES:
ICU stay | 30 days
  duration of stay in ICU

CONTACTS AND LOCATIONS:
Overall Officials: MATTEI Mathieu, MD, Principal Investigator — Central Hospital, Nancy, France
Locations (1):
- CHRU - Hopital de Brabois, Nancy, Lorraine, France

IPD SHARING:
Plan to Share IPD: Undecided